CLINICAL TRIAL: NCT05017272
Title: Technology Improving Success of Medication-Assisted Treatment in Primary Care - Phase 2
Brief Title: Technology for MAT in Primary Care - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Q2i, LLC (Industry)
Collaborators: University of California, Los Angeles (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-001516; 4R42DA050398-02 (NIH); 5R42DA050398-03 (NIH)
Record Dates: First submitted 2021-08-12; First posted 2021-08-23 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: Opioid use disorder; Primary care; mHealth; Medication for opioid use disorder; Technological solutions
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Using a "stepped wedge" effectiveness design, evaluate OARS platform in 6 treatment programs (N=200 treated patients) data before and after implementation along MAT outcomes. Each clinic, once randomized to begin using OARS, will have a minimum of 4 months and a maximum of 12 months to collect baseline data on the number of PCPs who have DATA-2000 waivers, on the number of patients each PCP treats and on relevant patient outcomes to MAT (e.g., length of time in treatment, visits kept with PCP and psychosocial providers, number of drug-free urine tests). There will be four months of baseline data available for PCPs and patients defined as treatment as usual (TAU) for clinics 1 and 2, eight months of baseline data available for PCPs and patients defined as TAU for clinics 3 and 4 and 12 months of baseline data available for PCPs and patients defined as TAU for clinics 5 and 6. In the final 3 months, we will finish data analyses, prepare papers for dissemination in peer-reviewed journals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Addiction Recovery Support (OARS) (Active Comparator): Data collected post-implementation of OARS in conjunction with medication for opioid use disorder (MOUD) at study sites.
  Interventions: Other: Opioid Addiction Recovery Support Software Platform
- Treatment as Usual (No Intervention): Data collected at baseline before OARS in conjunction with MOUD is implemented at study sites.

INTERVENTIONS:
Other: Opioid Addiction Recovery Support Software Platform — OARS (Opioid Addiction Recovery Support) is used by providers of MAT programs to improve insight into a patient's recovery progress while promoting ownership and adherence to treatment plans. OARS also provides extensive tools to support patients with recovery from Opioid Use Disorder.
  Other Names: OARS
  Arms: Opioid Addiction Recovery Support (OARS)

SUMMARY:
With over 72,000 overdose deaths in 2017, of which 47,600 are attributable to opioid overdose, the opioid epidemic has become North America's most widespread behavioral public health problem. Medication-assisted treatment (MAT) for opioid use disorder (OUD) is highly efficacious. The Opioid Addiction Recovery Support (OARS), comprised of a healthcare team portal connected to a patient mobile application, provides opioid-related education, promotes connectedness with clinicians, and tracks MAT treatment progress. This study will conduct interviews with patients that will inform optimal design of OARS, assess the efficacy of OARS in improving MAT outcomes in primary care settings, and evaluate the sustainability and return on investment.

It joins an outstanding scientific team at University of California, Los Angeles and a small business that has developed, Opioid Addiction Recovery Support (OARS) -- a software platform that by integrating with the Electronic Health Record (EHR) improves clinical management of patients by primary care providers (PCPs) treating patients with OUD using MAT. OARS platform uses a dashboard to show the real-time measurement of patient achievements in recovery. It provides opportunities for patients to interact with their PCPs, allowing for better connection to and support from their PCPs. OARS platform features artificial intelligence to analyze information from the EHR and from patients to provide a relapse risk assessment for patients receiving MAT for OUD, an innovation that sets OARS apart from other software solutions. The goal of Phase 1 was to modify the OARS platform for use in primary care settings by conducting interviews with Primary Care Physicians (PCPs) (N=20) and their patients with OUD (N=40) in primary care settings to collect data on feasibility and acceptability of engaging with OARS to inform the user-centered design of OARS.

The goals of Phase 2 of this study are to: (1) to assess the effectiveness of OARS in improving opioid agonist treatment outcomes across 6 treatment programs (N=200 treated patients) and (2) evaluate the sustainability and return on investment of OARS implementation across 6 treatment programs. A commercialization plan documents progress to date for the OARS platform and presents a market plan to improve both the scale and quality of MAT services delivered by PCPs in primary care, which is a major contribution to addressing the ongoing opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

* For Primary Care Providers (PCPs):

  * Physician, nurse practitioner, or physician's assistant in any area within primary care;
  * In possession of valid DATA-2000 waiver;
  * Currently treating more than two patients with OUD using oral buprenorphine-naloxone product;
  * Willing to distribute study materials to their patients describing the research and providing options for their participation.
* For Patient participants:

  * Diagnosed and treated using MAT within primary care setting (i.e., family medicine, internal medicine, adolescent medicine, pediatrics, obstetrics/gynecology, geriatrics, infectious diseases, emergency department, non-cancer pain management).

Exclusion Criteria:

* For PCPs:

  * Specialization outside primary care (e.g., psychiatry, neurology, etc) or provider works in specialized setting (e.g., addiction treatment programs; mental health clinic);
  * Not treating patients with OUD with oral buprenorphine-naloxone product (e.g., long-acting naltrexone or buprenorphine injections);
  * Individual interviews with physicians and their patients to discuss initially barriers and challenges to MAT for patients with OUD seen in primary care settings.
* For Patient participants:

  * MAT delivered in specialty care settings (i.e., psychiatry, substance abuse treatment programs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Behavioral and Addiction Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Further information about the OARS solution available here. — http://q2i.com/oars/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study utilized a non-randomized, stepped-wedge effectiveness trial design, which facilitates data collection on patient outcomes prior to the OARS intervention.
  Sites were purposefully selected and assigned to clusters as they were identified; one site in sequence 1, two sites in sequence 2, and one site in sequence 3.
  11 PCPs were enrolled in the study but only participated in semi-structured interviews to provide their insights on the OARS intervention.
Pre-assignment Details: Patient TAU baseline data (pre-intervention) were collected on patient outcomes retrospectively at the time of study enrollment. These baseline data were compared to corresponding data collected after OARS implementation (post-intervention) to determine the effectiveness of OARS. Data collection occurred through EHR data review and abstraction; no information was required directly from patients for the purpose of this study.
Units Other Than Participants: Clinics
Groups:
- Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention: Data collected pre- and post-implementation of OARS in conjunction with medication for opioid use disorder (MOUD) at the Wright Center study site.
- Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention: Data collected pre- and post-implementation of OARS in conjunction with medication for opioid use disorder (MOUD) at the Granville Vance and On-Call Mobile study sites.
- Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention: Data collected pre- and post-implementation of OARS in conjunction with medication for opioid use disorder (MOUD) at the Stallant Health study site.
Period: Step 1: Months 1-4
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started (All participants were on TAU during this period.) | 140; 1 Clinics | 3; 2 Clinics | 12; 1 Clinics
Completed | 140; 1 Clinics | 3; 2 Clinics | 12; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 2: Months 5-8
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started | 205; 1 Clinics (140 participants continued from TAU to start OARS and 65 new participants started OARS.) | 8; 2 Clinics (Months 5-7: 3 participants were in TAU, phase; Month 8: 3 participants from TAU started OARs and 5 new participants started OARs phase.) | 12; 1 Clinics
Completed | 205; 1 Clinics | 8; 2 Clinics | 12; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 3: Months 9-12
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started | 205; 1 Clinics | 8; 2 Clinics | 12; 1 Clinics
Completed | 205; 1 Clinics | 8; 2 Clinics | 12; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 4: Months 13-16
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started | 205; 1 Clinics | 8; 2 Clinics | 22; 1 Clinics (Month 13, 12 participants were still in TAU phase. Month 14-16: 12 participants from TAU phase started OARS and 10 new participants started OARs phase.)
Completed | 205; 1 Clinics (Stopped OARs at month 14.) | 8; 2 Clinics | 22; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 5: Months 17-20
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started | 0; 0 Clinics (Stopped OARs at month 14. No participants entered this period from this clinic.) | 8; 2 Clinics | 22; 1 Clinics
Completed | 0; 0 Clinics | 8; 2 Clinics (Stopped OARs at month 17.) | 22; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Step 6: Months 21-23
Arm/Group | Sequence 1: Months 1-4 TAU, Months 5-14 OARS Intervention | Sequence 2: Months 1-7 TAU, Months 8-17 OARS Intervention | Sequence 3: Months 1-13 TAU, Months 14-23 OARS Intervention
Started | 0; 0 Clinics (Stopped OARs at month 14. No participants entered this period from this clinic.) | 0; 0 Clinics (Stopped OARs at month 17. No participants entered this period from these two clinics.) | 22; 1 Clinics
Completed | 0; 0 Clinics | 0; 0 Clinics | 22; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: This study utilized a retrospective cohort-style, step-wedged trial design, which was based on cohort sampling (i.e., the same patients in each sequence were followed in each step from TAU to OARS). Patient Baseline Characteristic data were collected when participants started OARS.
  11 PCPs were enrolled in the study but only participated in semi-structured interviews to provide their insights on the OARS intervention. No other data was captured for PCPs.
Groups:
- Study Participants: All clinical trial participants.
Arm/Group | Study Participants
Number analyzed (Participants) | 235
Age, Continuous [Median (Full Range); unit: years] | 37 [32 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 147
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Non-Hispanic Black or African American | 10
  Non-Hispanic White | 212
  Non-Hispanic other race | 8
Region of Enrollment [Number; unit: participants]
  United States | 235

OUTCOME MEASURES:

1. Primary Outcome: Urine Drug Screening Test Results
Description: Percent of participants who had positive urine screening tests for buprenorphine, opioids (heroin, synthetics, fentanyl), cocaine, methamphetamine, benzodiazepines, cannabis.
  During the TAU period (pre-intervention), the percentage of all patient drug screens that were positive was calculated. The same was done during the OARS implementation period (post-intervention) for comparison with the TAU period (baseline).
Time Frame: Comparison of TAU baseline period (prior to start of intervention, up to 13 months) to OARS implementation period (start of intervention through to study completion, up to 10 months). Time Frames for the TAU and OARS periods differ by site.
Population: Reliable data for 80 participants during their TAU phase was not available.
Measure: Number; unit: percentage of participants positive
Groups:
- Treatment as Usual: Data collected at baseline before OARS in conjunction with MOUD is implemented at study sites. Reliable data for 80 participants during their TAU phase was not available.
Arm/Group | Opioid Addiction Recovery Support (OARS) | Treatment as Usual
Number analyzed (Participants) | 235 | 155
percentage of participants positive
  Buprenorphine | 92.3 | 92.0
  Opioids (heroin, synthetics, fentanyl) | 1.9 | 2.0
  Cocaine | 1.3 | 1.8
  Methamphetamine/Amphetamines | 0.9 | 2.0
  Benzodiazepines | 4.1 | 1.6
  Cannabis | 37.5 | 35.8

2. Primary Outcome: Appointment Attendance
Description: Percent of appointments scheduled and kept with Primary Care Provider.
  During the TAU period (pre-intervention), the percentage of attended appointments was calculated. The same was done during the OARS implementation period (post-intervention) for comparison with the TAU period (baseline).
Time Frame: as for outcome 1
Population: Reported percentages were calculated by dividing the number of attended appointments by total number of appointments (appointments attended + appointment no-shows).
  Reliable data for 80 participants during their TAU phase was not available.
Measure: Number; unit: percentage of appointments attended
Units Other Than Participants: Number of appointments
Arm/Group | Opioid Addiction Recovery Support (OARS) | Treatment as Usual
Number analyzed (Participants) | 235 | 155
Number analyzed (Number of appointments) | 4811 | 1539
percentage of appointments attended | 91.5 | 91.0

3. Secondary Outcome: OARS Features Use
Description: Type of OARS mobile phone app feature accessed by patient and level of patient involvement with each feature (times viewed per week).
  During the OARS implementation period (post-intervention), the type of OARS mobile phone app feature accessed by patient and level of patient involvement with each feature were calculated.
Time Frame: OARS implementation period (start of intervention through to study completion, up to 10 months). Time Frames for the OARS periods differ by site.
Population: Reliable data for 80 participants during their TAU phase was not available.
Measure: Median (Full Range); unit: times used per week
Arm/Group | Opioid Addiction Recovery Support (OARS)
Number analyzed (Participants) | 235
times used per week
  Viewed test results | 5 [0.0 to 7.5]
  Viewed progress | 1 [0.0 to 3.0]
  Viewed educational content | 1 [0.0 to 2.0]
  Sent chat message | 0 [0.0 to 3.0]
  Created journal entry | 0 [0.0 to 1.0]

4. Other Pre Specified Outcome: Return on Investment (ROI)
Description: ROI for a MAT provider using OARS compared to TAU.
  During the TAU period (pre-intervention), the ROI for MAT providers was calculated. The same was done during the OARS implementation period (post-intervention) for comparison with the TAU period (baseline).
Time Frame: as for outcome 1
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Counts of Services/Medications Received by Patients
Description: Including but not limited to visits, medications filled, reminder calls, asynchronous video related to OUD care.
  During the TAU period (pre-intervention), the counts of services/medications received by patients were determined. The same was done during the OARS implementation period (post-intervention) for comparison with the TAU period (baseline).
Time Frame: as for outcome 1
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Additional Healthcare Utilization by Patients
Description: Number of Emergency Department visits, Number of Medicaid charges, Number of inpatient stays, Number of other medications.
  During the TAU period (pre-intervention), healthcare utilization by patients was determined. The same was done during the OARS implementation period (post-intervention) for comparison with the TAU period (baseline).
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years.
Description: 11 PCPs were enrolled in the study but only participated in semi-structured interviews to provide their insights on the OARS intervention. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for PCPs.
Arm/Group | Opioid Addiction Recovery Support (OARS) | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/235 | 0/155
Other Adverse Events (participants affected / at risk) | 0/235 | 0/155

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic affected both enrollment and clinical operations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT05017272/Prot_SAP_000.pdf